CLINICAL TRIAL: NCT06778304
Title: A Randomized, Controlled, Open-label, Two-Period, Double-Crossover, Bioequivalence Clinical Trial: Comparing the Clinical Similarity of Recombinant Human Follicle-Stimulating Hormone JZB30 Injection With the Comparator Drug Gonal-f®
Brief Title: Bioequivalence Clinical Trial of Recombinant Human Follicle-stimulating Hormone JZB30
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Collaborators: Shanghai Jingze Biotechnology Co., Ltd. (Unknown); Chengdu Jingze pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yu Qin, Principal Investigator, West China Second University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: JZB30ART101
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Bioequivalence; Healthy Volunteers; Pharmacokinetics; Safety; Immunogenicity
Keywords: JZB30; Pharmacokinetics; Bioequivalence; Safety; Immunogenicity
MeSH Terms: interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants received a single subcutaneous injection of reference drug（Gonal F） (Active Comparator): On Day 1 (D1), participants received a single subcutaneous injection of the reference drug (injection site: 3-10 cm around the umbilical area) at a dose of 225 IU.
  Interventions: Drug: Gonal F
- participants received a single subcutaneous injection of test drug （JZB30） (Experimental): After a washout period of 8 to 10 days, the subjects entered the second period starting on Day 11 (D11) for crossover administration
  Interventions: Drug: jzb30

INTERVENTIONS:
Drug: Gonal F — The reference formulation is the recombinant human follicle-stimulating hormone injection (Gonal-f®) originally developed and produced by Merck Serono
  Other Names: Recombinant Human Follicle-stimulating Hormone
  Arms: participants received a single subcutaneous injection of reference drug（Gonal F）
Drug: jzb30 — The test formulation is the recombinant human follicle-stimulating hormone injection (code: JZB30) produced by Shanghai Jingze Biotechnology Co., Ltd./Chengdu Jingze Biopharmaceutical Co., Ltd.
  Other Names: Recombinant Human Follicle-stimulating Hormone
  Arms: participants received a single subcutaneous injection of test drug （JZB30）

SUMMARY:
Research Objective: Using the recombinant human follicle-stimulating hormone injection (Gonal-f®) originally developed by Merck Serono as the reference formulation, and the recombinant human follicle-stimulating hormone injection (code: JZB30) produced by Shanghai Jingze Biotechnology Co., Ltd./Chengdu Jingze Biopharmaceutical Co., Ltd. as the test formulation, a single-center, randomized, open-label, two-period, two-crossover designed bioequivalence study was conducted. The study aimed to evaluate the pharmacokinetic behavior, safety, and immunogenicity of the two formulations in healthy adult female Chinese subjects, providing a reference basis for rational clinical use.

DETAILED DESCRIPTION:
A total of 48 healthy adult female participants were enrolled. On Day 1 (D1), they received a single subcutaneous injection of either the test drug or the reference drug. After a washout period of 8 to 10 days, the subjects entered the second period starting on Day 11 (D11) for crossover administration. Pharmacokinetic (PK) blood samples were collected at specified time points, and the concentration of follicle-stimulating hormone (FSH) in the biological samples was measured using a validated electrochemiluminescence assay based on the MSD platform. The obtained PK data were used for pharmacokinetic analysis. Clinical safety assessments were conducted throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female participants aged 18-45 years (inclusive).
2. Body weight ≥45 kg, and body mass index (BMI) between 18-28 kg/m² (inclusive), where BMI = weight (kg) / height (m)².
3. Non-pregnant or non-lactating females.
4. Menstrual cycle length between 25-34 days (inclusive).
5. Females with a history of sexual activity but no plans for pregnancy.
6. Liquid-based/thin-layer cytology examination shows no clinically significant abnormalities.
7. Normal sex hormone levels, or abnormalities deemed clinically insignificant by the investigator.
8. Negative test results for HIV, HBV, HCV, or Treponema pallidum (T-trust).
9. Normal or clinically insignificant findings in medical history, physical examination, laboratory tests, and gynecological examinations (e.g., uterus and bilateral ovaries), as judged by the study physician.
10. Willing to participate in this clinical trial, understanding the study procedures, and able to provide written informed consent.

Subjects who do not meet any of the above criteria will not be eligible for participation as volunteers.

Exclusion Criteria:

1. Patients with polycystic ovary syndrome (PCOS).
2. Individuals with a history of FSH allergy, including those who have experienced ovarian hyperstimulation syndrome (OHSS) or are known to be allergic to gonadotropin-releasing hormone agonists (GnRH-a) or their analogs.
3. Individuals with special dietary requirements during hospitalization who cannot adhere to a standardized diet.
4. Individuals with a medical history of ovarian, breast, uterine, hypothalamic, or pituitary diseases deemed clinically significant by the investigator, or a history of thrombosis or current thrombotic disorders.
5. Individuals with diminished ovarian reserve.
6. Individuals engaged in intense physical activities, such as professional athletes.
7. Individuals who have used any prescription drugs or therapeutic medications within 1 week prior to dosing.
8. Individuals using hormonal contraceptives (short-term contraceptives within 3 months before screening or long-term contraceptives within 6 months before screening).
9. Individuals with alcohol abuse (defined as consuming more than 21 standard units of alcohol per week, where 1 standard unit contains 14 g of alcohol, e.g., 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine) or frequent alcohol consumption within 6 months before screening (defined as consuming more than 14 standard units per week, e.g., 240 mL of beer, 30 mL of 40% spirits, or 100 mL of wine) or alcohol consumption within 24 hours before dosing.
10. Individuals who are heavy smokers (smoking more than 5 cigarettes per day within 3 months before the trial) or cannot comply with the smoking ban during the trial.
11. Individuals with a history of drug abuse (e.g., morphine, methamphetamine, ketamine, MDMA, THC, etc.).
12. Individuals who consume strong coffee or tea daily.
13. Individuals who have donated blood or experienced blood loss ≥400 mL within 3 months.
14. Individuals who have participated in any drug clinical trial as a subject within 3 months before this trial.
15. Individuals deemed unsuitable for participation by the investigator.

Exclusion:

Subjects who meet any of the above criteria will not be eligible for participation.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) | First Period: From pre-dose (0 hour) to 168 hours post-dose on Day 1 (D1). Second Period: From pre-dose (0 hour) to 168 hours post-dose on Day 11 (D11)
  To evaluate the bioequivalence between the test formulation (JZB30) and the reference formulation (Gonal-f®) by comparing their pharmacokinetic parameters, including AUC (area under the curve), Cmax (maximum plasma concentration), and Tmax (time to reach maximum concentration), in healthy adult female subjects.
Cmax (maximum plasma concentration) | First Period: From pre-dose (0 hour) to 168 hours post-dose on Day 1 (D1). Second Period: From pre-dose (0 hour) to 168 hours post-dose on Day 11 (D11)
  To evaluate the bioequivalence between the test formulation (JZB30) and the reference formulation (Gonal-f®) by comparing their pharmacokinetic parameters, including AUC (area under the curve), Cmax (maximum plasma concentration), and Tmax (time to reach maximum concentration), in healthy adult female subjects.

SECONDARY OUTCOMES:
ADA（Anti-Drug Antibodies） | First Period: Pre-dose (0 hour) and 168 hours post-dose on Day 1 (D1). Second Period: Pre-dose (0 hour) and 168 hours post-dose on Day 11 (D11). Follow-up: Up to 7 days after the last dose in the second period (Day 18).
  To evaluate the immunogenicity of the test formulation (JZB30) and the reference formulation (Gonal-f®) by detecting the presence of anti-drug antibodies (ADA) and assessing their potential impact on pharmacokinetics and safety in healthy adult female subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Principal Investigator — National Drug Clinical Trial Institution of West China Second Hospital
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Chen Z, Yu Q, Feng S, Mo L, Cai L, Du C, Du D, Zou Q. A single-center, randomized, open-label, two-period, crossover, fasted bioequivalence study: comparing recombinant human follicle-stimulating hormone for injection (JZB30) with Gonal-f(R) in healthy Chinese female participants. Front Pharmacol. 2025 Nov 10;16:1678830. doi: 10.3389/fphar.2025.1678830. eCollection 2025. PMID 41293254